CLINICAL TRIAL: NCT00211965
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blinded Study to Evaluate Safety and Immunogenicity of StaphVAX®, a Bivalent Staphylococcus Aureus Glycoconjugate Vaccine in Adult Patients Receiving an Orthopedic Prosthetic Implant
Brief Title: StaphVAX Immunogenicity and Safety in Orthopaedic Joint Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Collaborators: Public Health England (Other Government)
Responsible Party: Matt Hohenboken, MD, PhD, Executive Director Clinical & Medical Affairs, Nabi Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nabi-1363
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Staphylococcal Infections
Keywords: Knee replacement surgery; hip replacement surgery; nosocomial infections; Arthroplasty
MeSH Terms: conditions — Staphylococcal Infections; Cross Infection | interventions — StaphVax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vaccine (Experimental): single dose
  Interventions: Biological: S. aureus Types 5 and 8 Capsular Polysaccharide Conjugate
- placebo (Placebo Comparator): single dose
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: S. aureus Types 5 and 8 Capsular Polysaccharide Conjugate — single IM dose of 200 mcg total conjugate
  Other Names: StaphVAX®
  Arms: vaccine
Biological: placebo — single dose IM
  Arms: placebo

SUMMARY:
Staphylococcus aureus (S. aureus) is the most common pathogen encountered in infections associated with orthopedic surgery. StaphVAX® is a bivalent S. aureus types 5 and 8 vaccine which contains the purified capsular polysaccharides that have been implicated as a major factor in the invasiveness of S. aureus. Immunoprophylaxis by vaccinating against S. aureus prior to surgery could provide sufficient antibody concentrations during surgery and the wound healing period so as to decrease the risk of S. aureus infection. This study aims to demonstrate the immunogenicity and safety of a single dose of StaphVAX in patients who are candidates for orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Candidate for knee or hip replacement
* Expectation of protocol compliance
* Negative pregnancy test, where appropriate

Exclusion Criteria:

* Known S. aureus infection in the prior 3 months
* Infection in the prior 2 weeks
* Known HIV infection
* Immunomodulatory drugs
* Malignancy (other than basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, or early prostate cancer)
* Hypersensitivity to components of StaphVAX

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-04; Primary Completion 2006-05 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Sero-type specific antibody concentrations | 6 weeks after study dose

SECONDARY OUTCOMES:
Sero-type specific antibody concentrations | various other time points after study dose, up to 26 wk
adverse events | throughout 6 months observation after study dose

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hohenboken, MD, PhD, Study Director — Nabi Biopharmaceuticals
Locations (1):
- National Royal Orthopaedic Hospital, Stanmore, Middlesex, United Kingdom